CLINICAL TRIAL: NCT01169974
Title: Evaluation Chez Des Sujets Volontaires Sains de l'ischémie-reperfusion cutanée
Brief Title: Use of Laser Speckle to Study Post Occlusive Reactive Hyperhemia in Healthy Subjects
Acronym: SpeckleShake
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: CHU P 2010-18
Record Dates: First submitted 2010-07-23; First posted 2010-07-26 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Microcirculation
Keywords: Microcirculation; laser flowmetry; Skin; Physiology
MeSH Terms: interventions — Laser-Doppler Flowmetry; Blood Gas Monitoring, Transcutaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- healthy volunteers
  Interventions: Other: tourniquet ischemia

INTERVENTIONS:
Other: tourniquet ischemia — Recording of cutaneous blood flow on the forearm at rest before and following tourniquet ischemias of 1 , 2 & 3 minutes
  Other Names: Laser doppler flowmetry; Transcutaneous oxygen pressure; Near infra-red spectrometry; Plethysmography

SUMMARY:
The investigators aim to test the hypothesis that Laser speckle contrast imaging allows for the measurement of cutaneous blood flow following various durations of tourniquet ischemia.

DETAILED DESCRIPTION:
Ischemia and post occlusive reactive hyperemia in the skin is tested in healthy normal subjects for tourniquet ischemias of 1, 2 & 3 minutes at rest.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Affiliation to the French health system

Exclusion Criteria:

* Any disease or chronic treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2011-02-01 (Actual); Primary Completion 2012-09 (Actual); Study Completion 2012-12-04 (Actual)

PRIMARY OUTCOMES:
Laser speckle | with 2 minutes of ischemia
  Peak value of laser speckle signal

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Mahe, Principal Investigator — University Hospital in Angers
Locations (1):
- University hospital, Angers, France